CLINICAL TRIAL: NCT06693687
Title: A Study of the ApricityCare Program for Early Detection and Management of Treatment-Related Adverse Events in Patients With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0229; NCI-2024-09566 (Other: NCI-CTRP Clinical Trials Registry])
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic Cancer (Other): Participants will have 24/7 access to the ApricityCare service. Participants can check in and report any symptoms or side effects through the ApricityCare app, or by phone, at any time.
  Participants will be asked to report your status at least weekly, even if participants are not experiencing any side effects. ApricityCare nurses will review each participants report and provide appropriate education and/or virtual management or escalate, as needed, to the study doctor or emergency service, based on guidelines. Each encounter with an ApricityCare nurse will be sent to the electronic health record (EHR) in real time for review/inclusion into your medical record.
  For any in-person visits participants attend, the study doctor will review the ApricityCare symptom summary with participants. For all these visits, please bring your smartphone, which carries the ApricityCare application, for this review.
  Interventions: Behavioral: Metastatic Cancer

INTERVENTIONS:
Behavioral: Metastatic Cancer — Participants will be asked to to take part in a research study because you have metastatic cancer (meaning that your cancer has spread to other parts of the body) and will be starting systemic therapy.

SUMMARY:
To evaluate the rate of therapy discontinuation due to toxicity (side effects) among participants with cancer using ApricityCare.

Investigators want to learn if identification of early clinical signs of irAEs with timely treatment can prevent severity progression and reduce treatment discontinuation.

DETAILED DESCRIPTION:
Primary Objective • To determine the rate of therapy discontinuation due to toxicity among patients using ApricityCare.

Secondary Objectives

• To evaluate time the ease and experience of patient use of ApricityCare (i.e., patient engagement) in reporting symptoms during their systemic cancer treatments. Furthermore, the frequency of patient symptom reporting via check-in to ApricityCare will be evaluated, as will the time taken to respond and engage patients after they report toxicity or other adverse events via ApricityCare.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Confirmed diagnosis of cancer

  * Part 1 (Run-in Phase): Only patients with prostate, kidney, and/or bladder cancer will be enrolled with either localized or metastatic disease.
  * Part 2 (Expansion Phase): Metastatic patients will be enrolled. Note, evaluable metastatic patients from Ppart 1 will be counted in Cohort A as described in section 8.4.
* Planned to receive systemic anti-cancer therapy
* Ability to understand and the willingness to sign a written informed consent document
* Ability to speak, read, and understand one of the following languages: English, Spanish, Mandarin and Cantonese Chinese
* Ownership of a smartphone and willingness to use it as outlined by the protocol and described in the ICF

Exclusion Criteria:

- Have any medical, psychological, or social condition that, in the opinion of the investigator would preclude participation in this study (pregnancy is not exclusionary and pregnant women will be permitted to enroll in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org